CLINICAL TRIAL: NCT01916759
Title: Systems Biological Responses to Influenza Vaccination in an HIV-infected and HIV-uninfected Adult Population in Kampala, Uganda
Brief Title: Differences in Response to the Flu Vaccine Among Adults With HIV and Without HIV in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Saad B. Omer, PhD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00058919; 1U19AI090023-02 (NIH)
Record Dates: First submitted 2013-02-25; First posted 2013-08-06 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome; Influenza
Keywords: immunization
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIV uninfected adults (Other): 25 HIV uninfected adults enrolled at the Mulago National Referral Hospital complex in Kampala, Uganda will receive seasonal trivalent inactivated influenza vaccine (Vaxigrip®).
  Interventions: Drug: Seasonal trivalent inactivated influenza vaccine (Vaxigrip®)
- HIV infected adults on HAART (Other): 25 HIV infected adults enrolled at the Mulago National Referral Hospital complex in Kampala, Uganda will receive seasonal trivalent inactivated influenza vaccine (Vaxigrip®).
  Interventions: Drug: Seasonal trivalent inactivated influenza vaccine (Vaxigrip®)
- HIV-infected long-term non-progressors (Other): 10 HIV-infected long-term non-progressor adults enrolled at the Mulago National Referral Hospital complex in Kampala, Uganda will receive seasonal trivalent inactivated influenza vaccine (Vaxigrip®).
  Interventions: Drug: Seasonal trivalent inactivated influenza vaccine (Vaxigrip®)

INTERVENTIONS:
Drug: Seasonal trivalent inactivated influenza vaccine (Vaxigrip®) — Administer seasonal trivalent inactivated influenza vaccine (Vaxigrip®) and collect blood specimens at 0, 1, 3, 7, 14, 28 and 100 days following vaccination.

SUMMARY:
To use a systems biological approach to study the molecular signatures of innate and adaptive responses to vaccination in a HIV infected versus uninfected adult population in Kampala, Uganda.

DETAILED DESCRIPTION:
This longitudinal, observational cohort study will be conducted at the Makerere University- Johns Hopkins University Research Collaboration, at the Mulago National Referral Hospital complex in Kampala Uganda. The study will consist of 2 groups. One group will consist of 25 healthy HIV uninfected adults and the other arm will consist of 35 HIV infected adults. Within the HIV infected arm there will be two groups, 25 HIV infected adults and 10 long term non-progressors. Vaccinees will receive a primary immunization at day 0, and blood samples will be obtained at days 0, 1, 3, 7, 14, 28 and 100 after immunization.

We will analyze the early molecular signatures (identified by microarray analyses, as well as by FACS analyses of innate immune cells and luminex analyses of cytokines and chemokines) that correlate and predict the later immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. For HIV uninfected group

   * Confirmation of HIV-1 infection from medical records
2. For HIV infected on HAART group

   * Confirmation of HIV-1 infection from medical records
   * Participants must be on HAART for at least 6 months prior to enrollment
   * A CD4 T-cell count available in the last 6 months
   * CD4 T-cell count >350 cells/μL on the eligibility blood specimen
3. Long-term non-progressor group

   * HIV infected for more than 7 years
   * No evidence of opportunistic infections in the medical records
   * Never received antiretroviral therapy (except anti-retrovirals for prevention of mother-to-infant transmission of HIV)
   * A CD4 T-cell count available in the last 6 months
   * CD4+ T-cell count slop of ≥0 cells/µl blood from entry into the MU-JHU cohort until the most recent available CD4+ T-cell count.

Exclusion Criteria:

1. Current moderate or severe acute illness, history of fever or temperature ≥37.5oC within 48 hours prior to vaccination (participants can be re-evaluated at a subsequent visit)
2. History of systemic disease, including: Guillain-Barré Syndrome; known hepatitis B, or hepatitis C infection; cardiac disease; uncontrolled diabetes mellitus (including gestational diabetes); chronic liver condition; clinically significant renal impairment; clinically significant neurological disorders; active TB within the last year; Cancer. This information will be based on self-reporting and (where possible) will be confirmed by hospital medical records
3. Received immunoglobulin or other blood product within the preceding 3 months or expected receipt of blood products during the 3 months of follow-up
4. History of anaphylactic hypersensitivity reactions to egg proteins (eggs or egg products), or any other component of the vaccine including traces (formaldehyde, octoxinol 9 (Triton X-100) and neomycin)
5. History of severe reaction (including hypersensitivity) after receiving any vaccine
6. Currently pregnant
7. In the opinion of the study team it would be unsuitable for the study subjects to receive the vaccine or participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
In group and between group comparison of immune parameters and gene expressions that change significantly following vaccination with the seasonal trivalent influenza vaccine (Vaxigrip®) | From baseline (Day 0) to 100 days post vaccination
  Immune parameters or gene expressions that change significantly in groups over baseline post immunization and between the study groups will be analyzed. For immune parameters, we will use a two-sided paired t-test. Fold-change will be combined with the test p-value in a selection criterion as appropriate. The tentative selection criterion is p-value ≤ 0.01 and fold change ≥ 3. For the gene/miRNA expression data, we will use the method Significance Analysis of Microarrays (SAM) with paired design to find differentially expressed genes. False discovery rate (FDR) will be used as selection criterion. The tentative selection criterion is FDR ≤ 0.1.
Proportion of subjects achieving 4-fold or greater hemagglutination inhibition (HAI)antibody titer increases. | From baseline (Day 0) to 100 days following primary vaccination
  Proportion of subjects in different study groups achieving 4-fold or greater hemagglutination inhibition (HAI)antibody titer increases will be tabulated at each time point (Days 0, 1, 3, 7, 14, 28 and 100) and plotted across time. Fisher's exact test will be used to make comparisons between the study groups.
Calculating correlation coefficient between the immune parameter and vaccine immunogenicity, as measured by the humoral immune response against seasonal influenza. | From baseline (Day 0) to 100 days post vaccination
  For immune parameters, we will calculate the correlation coefficient between the immune parameter and vaccine immunogenicity, as measured by the humoral immune response against seasonal influenza. The p-values associated with the correlation coefficients will be used to select immune parameters that are associated with the respective adaptive immune responses. The tentative selection criterion is p-value ≤ 0.01. For gene expression data, we will use the method Significance Analysis of Microarrays (SAM) with quantitative outcome to identify genes that are significantly associated with the immune response. False discovery rate (FDR) will be used as selection criterion. The tentative selection criterion is FDR ≤ 0.1.
Characterization of the gut microbiota to determine compositional differences between HIV-uninfected adults versus HIV-infected adults on HAART versus HIV-infected long-term non-progressors | From baseline (Day 0) to Day 28 post vaccination
  Gut mircobiota will be characterized to determine what compositional differences exist between HIV-uninfected adults versus HIV-infected adults on HAARt versus HIV-infected long-term non-progressors at baseline (Day 0), Day 7 and Day 28 post vaccination
Correlation between microbiata status and the quality of immune response elicited in vaccinated individuals | From baseline (Day 0) to Day 28 post vaccination
  Determine whether the status of the microbita correlates with the quality of immune responses elicited in vaccinated individuals

CONTACTS AND LOCATIONS:
Overall Officials: Saad B Omer, MBBS,MPH,PhD, Principal Investigator — Emory Unversity
Locations (1):
- Makere University- Johns Hopkins University Research Collaboration, at the Mulago National Referral Hospital, Kampala, Uganda

REFERENCES:
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Nakaya HI, Wrammert J, Lee EK, Racioppi L, Marie-Kunze S, Haining WN, Means AR, Kasturi SP, Khan N, Li GM, McCausland M, Kanchan V, Kokko KE, Li S, Elbein R, Mehta AK, Aderem A, Subbarao K, Ahmed R, Pulendran B. Systems biology of vaccination for seasonal influenza in humans. Nat Immunol. 2011 Jul 10;12(8):786-95. doi: 10.1038/ni.2067. PMID 21743478
- [Background] Beck JM, Rosen MJ, Peavy HH. Pulmonary complications of HIV infection. Report of the Fourth NHLBI Workshop. Am J Respir Crit Care Med. 2001 Dec 1;164(11):2120-6. doi: 10.1164/ajrccm.164.11.2102047. No abstract available. PMID 11739145
- [Background] Malaspina A, Moir S, Orsega SM, Vasquez J, Miller NJ, Donoghue ET, Kottilil S, Gezmu M, Follmann D, Vodeiko GM, Levandowski RA, Mican JM, Fauci AS. Compromised B cell responses to influenza vaccination in HIV-infected individuals. J Infect Dis. 2005 May 1;191(9):1442-50. doi: 10.1086/429298. Epub 2005 Mar 24. PMID 15809902
- [Background] Zanetti AR, Amendola A, Besana S, Boschini A, Tanzi E. Safety and immunogenicity of influenza vaccination in individuals infected with HIV. Vaccine. 2002 Dec 20;20 Suppl 5:B29-32. doi: 10.1016/s0264-410x(02)00511-x. PMID 12477415
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Tebas P, Frank I, Lewis M, Quinn J, Zifchak L, Thomas A, Kenney T, Kappes R, Wagner W, Maffei K, Sullivan K; Center for AIDS Research and Clinical Trials Unit of the University of Pennsylvania. Poor immunogenicity of the H1N1 2009 vaccine in well controlled HIV-infected individuals. AIDS. 2010 Sep 10;24(14):2187-92. doi: 10.1097/QAD.0b013e32833c6d5c. PMID 20616698
- [Background] Pallikkuth S, Kanthikeel SP, Silva SY, Fischl M, Pahwa R, Pahwa S. Innate immune defects correlate with failure of antibody responses to H1N1/09 vaccine in HIV-infected patients. J Allergy Clin Immunol. 2011 Dec;128(6):1279-85. doi: 10.1016/j.jaci.2011.05.033. Epub 2011 Jul 12. PMID 21752440
- [Background] Wrammert J, Smith K, Miller J, Langley WA, Kokko K, Larsen C, Zheng NY, Mays I, Garman L, Helms C, James J, Air GM, Capra JD, Ahmed R, Wilson PC. Rapid cloning of high-affinity human monoclonal antibodies against influenza virus. Nature. 2008 May 29;453(7195):667-71. doi: 10.1038/nature06890. Epub 2008 Apr 30. PMID 18449194
- [Background] Wrammert J, Koutsonanos D, Li GM, Edupuganti S, Sui J, Morrissey M, McCausland M, Skountzou I, Hornig M, Lipkin WI, Mehta A, Razavi B, Del Rio C, Zheng NY, Lee JH, Huang M, Ali Z, Kaur K, Andrews S, Amara RR, Wang Y, Das SR, O'Donnell CD, Yewdell JW, Subbarao K, Marasco WA, Mulligan MJ, Compans R, Ahmed R, Wilson PC. Broadly cross-reactive antibodies dominate the human B cell response against 2009 pandemic H1N1 influenza virus infection. J Exp Med. 2011 Jan 17;208(1):181-93. doi: 10.1084/jem.20101352. Epub 2011 Jan 10. PMID 21220454
- [Background] Morita R, Schmitt N, Bentebibel SE, Ranganathan R, Bourdery L, Zurawski G, Foucat E, Dullaers M, Oh S, Sabzghabaei N, Lavecchio EM, Punaro M, Pascual V, Banchereau J, Ueno H. Human blood CXCR5(+)CD4(+) T cells are counterparts of T follicular cells and contain specific subsets that differentially support antibody secretion. Immunity. 2011 Jan 28;34(1):108-21. doi: 10.1016/j.immuni.2010.12.012. Epub 2011 Jan 6. PMID 21215658
- [Background] DAIDS table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004, Clarification August 2009. Available at rcc.tech-res-intl.com.